CLINICAL TRIAL: NCT00003666
Title: Phase II Trial of 6-Hydroxymethylacylfulvene (HMAF; MGI-114) in Patients With Relapsed or Refractory Non-Small Cell Lung Cancer
Brief Title: Irofulven in Treating Patients With Relapsed or Refractory Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39805; U10CA031946 (NIH); CLB-39805; CDR0000066761 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HMAF (Experimental): treatment of refractory or relapsed NSCLC with HMAF
  Interventions: Drug: 6-hydroxymethylacylfulvene

INTERVENTIONS:
Drug: 6-hydroxymethylacylfulvene — 11mg/sq m IV infusion over 5 min q day for 5 days each 28 day cycle
  Other Names: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients with relapsed or refractory non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate to 6-hydroxymethylacylfulvene (HMAF) as salvage chemotherapy in patients with relapsed or refractory non-small cell lung cancer. II. Determine the duration of response to this regimen in this patient population. III. Determine the effect of prior response to chemotherapy on the response to HMAF in these patients. IV. Determine the survival and failure-free survival of patients treated with HMAF. V. Evaluate the toxicity profile of HMAF as salvage therapy in these patients.

OUTLINE: Patients are stratified into relapsed or refractory patient groups based on results achieved with prior therapy. Patients receive 6-hydroxymethylacylfulvene IV over 5 minutes daily for 5 days. Courses repeat every 28 days. Patients with stable or responding disease are treated for a minimum of 6 courses (2 courses beyond optimal response) in the absence of unacceptable toxic effects or disease progression. Patients are followed at least every 3 months for 1 year, then every 6 months until death.

PROJECTED ACCRUAL: A total of 66 patients (33 for each stratum) will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven recurrent or refractory non-small cell lung cancer Squamous cell Adenocarcinoma (including bronchoalveolar cell) Large cell anaplastic (giant and clear cell carcinomas) Measurable disease (not bone disease only, pleural or pericardial effusions, or irradiated lesions, unless progression is documented after radiotherapy) No CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater 1.5 mg/dL SGOT no greater than 2 times upper limit of normal (ULN) Renal: Creatinine no greater than ULN Cardiovascular: No active cardiac disease No unstable angina No myocardial infarction within 6 months No congestive heart failure No inability to tolerate hypotension Other: Not pregnant or nursing Fertile patients must use effective contraception HIV negative No uncontrolled diabetes mellitus No psychiatric disorders No concurrent secondary malignancies except nonmelanomatous skin cancer or patients with less than a 30% risk of relapse

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since mitomycin) At least 1 prior chemotherapy agent or combination, including adjuvant or neoadjuvant therapy for non-small cell lung cancer No more than 1 prior chemotherapy agent or combination for metastatic or recurrent disease No prior HMAF No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy except for nondisease related conditions Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No concurrent palliative radiotherapy Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 1998-11; Primary Completion 2004-09 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Response | ea tx cycle; q 3 mon Yr 1 post tx, then q 6 mon until progression

SECONDARY OUTCOMES:
Toxicity | Each tx cycle

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Sherman, MD, Study Chair — Medical University of South Carolina
Locations (48):
- United States (48):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Veterans Affairs Medical Center - Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Sherman CA, Herndon JE 2nd, Watson DM, Green MR; Cancer and Leukemia Group B. A phase II trial of 6-hydroxymethylacylfulvene (MGI-114, irofulven) in patients with relapsed or refractory non-small cell lung cancer. Lung Cancer. 2004 Sep;45(3):387-92. doi: 10.1016/j.lungcan.2004.02.017. PMID 15301880
- [Result] Sherman CA, Herndon JE, Green MR, et al.: CALGB 39805: phase II trial of 6-hydroxymethylacylfulvene (HMAF; MGI-114) in patients with relapsed or refractory non-small cell lung cancer (NSCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 19: A2163, 2000.